CLINICAL TRIAL: NCT02943720
Title: A Multicentre, Double-blind, Placebo-Controlled, Randomized Trial to Assess the Efficacy and Tolerability of Two Dosing Regimens of AllerT in Adults With Birch Pollen Allergic Rhinitis
Brief Title: ATIBAR - Efficacy and Safety of Two Doses of AllerT in Patients Allergic to Birch Pollen
Acronym: ATIBAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anergis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN006T
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): 5 SC injections in 2 months
  Interventions: Drug: placebo
- AllerT 50 ug (Experimental): 5 SC injections in 2 months
  Interventions: Drug: AllerT
- AllerT 10 ug (Experimental): 5 SC injections in 2 months
  Interventions: Drug: AllerT

INTERVENTIONS:
Drug: AllerT — Bet v 1 contiguous overlapping peptides mixed with aluminium hydroxide solution
  Arms: AllerT 10 ug; AllerT 50 ug
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
A multicentre, Double-blind, Placebo-Controlled, Randomized Trial to Assess the Efficacy and Tolerability of Two Dosing Regimens of AllerT, a Combination of Contiguous Overlapping Peptides Derived from Bet v 1, in Adults with Birch Pollen Allergic Rhinitis/Rhinoconjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 to 65 yrs old, male or female
* moderate to severe allergic Rhinitis/Rhinoconjunctivitis to birch pollen during the two preceding birch pollen seasons
* positive Skin Prick Test (SPT) to birch pollen extract
* positive specific IgE CAP to Bet v1.

Exclusion Criteria:

* persistent non-controlled asthma (Forced Expiratory Volume, FEV1 < 85% of predicted),
* previous specific immunotherapy (SIT) to tree pollens,
* previous SIT to any allergen within 5 years,
* previous history of severe anaphylactic reaction,
* perennial allergic Rhinitis/Rhinoconjunctivitis,
* other disorder possibly influencing the trial outcomes,
* pregnancy,
* any severely debilitating disease,
* primary or secondary immunodeficiency or treatment with immunosuppressor drugs within one month prior to randomization (oral steroids, other immunosuppressors).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Combined Symptom and Medication Score (CSMS) | 2 to 6 months after the end of treatment
  the CSMS will be assessed daily throughout the first birch pollen season following the end of the preseasonal 2-month treatment. The difference in average daily CSMS per treatment group will be compared taking into account all days of the birch pollen season at each study center. All patients will receive treatment during the preceding winter or spring and will thus have the primary outcome assessment performed between 2 and 6 months after the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Durham, MD, Study Chair — NHLI, Imperial College London
Locations (36):
- Denmark (5):
  - Lungemedicinsk Forskningsafdeling,, Aarhus
  - Herlev-Gentofte Hospital, Hud - og Allergiafdelingen,, Hellerup
  - Kolding Hospital, Kolding
  - Næstved Sygehus, Lungemedicinsk avd, Næstved
  - Odense Universitetshospital, Odense
- Finland (2):
  - Oulun Yliopistollinen sairaala Korva-, nenä- ja kurkkutautien poliklinikka., Oulu
  - TYKS T-sairaala Allergiayksikkö TA2, Turku
- Germany (7):
  - HNO Heilkunde u. Allergologie praxis, Berlin
  - HNO Praxis Dr Yarin, Dresden
  - HNO Praxis Dr Thieme, Duisburg
  - HNO Praxis Dr Horn, Heidelberg
  - Dres Heimlich HNO praxis, Heidelberg
  - Medamed, Leipzig
  - Zentrum fur Rhinologie une Allergologie, Wiesbaden
- Lithuania (4):
  - Hospital of Lithuanian University, Kaunas
  - CD8 Klinika, Kaunas
  - Vilnius University Hospital, Vilnius
  - Vilnius City Clinical hospital, Vilnius
- Norway (3):
  - Harestua Medisinske Senter, Harestua
  - KAL Kliniken, Oslo
  - Ski Ore-Nese-Hals, Ski
- Poland (7):
  - Clinica Vitae, Gdansk
  - Grazyna Pulka Specjalistyczny Osradek All-Med, Krakow
  - Malopolskie Centrum Alergologii, Krakow
  - EMED Centrum Uslug Medycznych, Rzeszów
  - Clinmedica Research OMC, Skierniewice
  - All-Med Specjalistyczna Opieka Medyczna, Wroclaw
  - NZOZ-ALER-med Specjalistyczna Opieka Medycna, Wroclaw
- Slovakia (7):
  - ALIAN s.r.o. Ambulancia alergologie, Bardejov
  - Imunologia a alergologia, Komárno
  - ALERSA s.r.o. Imunoalergologicka ambulancia, Košice
  - STALERG s.r.o. Imunoalergologicka ambulancia, Košice
  - DANIMED s.r.o. Ambulancia klinickejimunologie a alergologie, Levice
  - EMED s.r.o. Alergoimunologické centrum, Prešov
  - Imunoalergologicka ambulancia, Šurany
- Karolinska Trial Alliance, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided